CLINICAL TRIAL: NCT04179097
Title: Dichrotic Notch Positioning in Finger Photoplethysmography Waveform Reflex Systemic Vascular Resistance
Brief Title: Photoplethysmographic Dichrotic Notch Reflexes Systemic Hemodynamics
Status: Terminated | Type: Observational
Why Stopped: COVID pandemic changed completely the surgical schedule and human resources in our hospital. It was impossible to coordinate the anesthesiologists involved in the study with the kind of patients need for this particular study.
Sponsor: Hospital Privado de Comunidad de Mar del Plata (Other)
Responsible Party: Sponsor
Other Study IDs: 2919/1942/2019
Record Dates: First submitted 2019-09-30; First posted 2019-11-26 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Vascular Diseases
Keywords: Doppler; Photoplethysmography
MeSH Terms: conditions — Vascular Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Finger photoplethysmography — Bilateral finger photoplethysmogray, bilateral brachial artery Doppler, Aorta artery Doppler
  Other Names: Brachial and aorta Doppler

SUMMARY:
Changes in the vascular tone of anesthetized patients is common and cause hemodynamic problems. The investigators have previously demonstrated that the shape of the pulse oximetry waveform (photoplethysmography) is closely related to the changes observed in systemic vascular resistence. The main change in pulse waveform is based to the dichrotic notch position. The present study was designed to determine if the dichrotic notch position is related to a local or a systemic change in the vascular tone.

DETAILED DESCRIPTION:
This is a prospective and observational study designed to determine if the changes observed in finger photoplethysmographic waveform of surgical patients is related to a local or a sistemic changes in the vascular tone. The investigators will studied 15 patients undergoing regional brachial plexus anesthesia for upper limb surgeries. Photoplethysmography will be continuously recorded in the thumb of the tested hand (anesthetized hand) and in the thumb of the control, opposite hand. Duplex color and power Doppler will measure flow in the both brachial arteries and in the aorta (supraesternal view). The contour analysis of both, photoplethysmogram and arterial flow velocities will be analyzed, correlated and compared.

ELIGIBILITY:
Inclusion Criteria:

* Written Inform Consent
* Programmed surgery
* Supine position

Exclusion Criteria:

* Emergency surgery
* Peripheral vascular diseases

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients undergoing regional anesthesia (brachial plexus block) for upper limb surgeries
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2019-11-05 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-10 (Actual)

PRIMARY OUTCOMES:
Analysis in the position of the dichrotic notch between photoplethysmogram and spectral Doppler waveforms. | 4 hours
  The position of the dichrotic notch of pulse waveform in photoplethysmogram (time arrival of diastolic wave expressed in seconds) was compared to the one observed in the spectral Doppler waveform (seconds).

CONTACTS AND LOCATIONS:
Overall Officials: Gerardo Tusman, MD, Principal Investigator — Hospital Privado de Comunidad
Locations (2):
- Argentina (2):
  - Cecilia M. Acosta, Mar del Plata, Buenos Aires
  - Hospital Privado de Comunidad, Mar del Plata, Buenos Aires

IPD SHARING:
Plan to Share IPD: No